CLINICAL TRIAL: NCT00548795
Title: A Prospective Assessment of Viral-induced Adaptation of Neutrophil Response in ARDS - Ancillary to ARDS Network Trials
Brief Title: Viral-Related Neutrophil Response and Condition Severity in People With ARDS
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jerry A. Nick, M.D., Principal Investigator, National Jewish Health
Other Study IDs: 1424; R01HL090991 (NIH)
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute Respiratory Distress Syndrome; ARDS; Neutrophil
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a severe lung condition that can result from a bacterial infection in the lungs. Viral infections may impair the body's immune system response to bacteria, which may lead to more serious lung injury. This study will evaluate the association between the immune response and ARDS severity in people who have ARDS plus a viral infection.

DETAILED DESCRIPTION:
ARDS is a serious condition that involves inflammation and fluid accumulation in the lungs, leading to low blood oxygen levels and breathing failure. It is often fatal and affects approximately 150,000 individuals each year in the United States. Common underlying causes include bacterial infections, lung trauma, and pneumonia. Even in people with similar risk factors for ARDS, there are often varying levels of condition severity. This may be because some people experience an ongoing viral infection that further predisposes them to the bacterial infection, worsening the severity of ARDS. Viruses release a protein called Type I interferon. This protein increases the response of the interferon stimulated genes (ISG) in neutrophils, which are white blood cells that protect the body against disease and infections by destroying bacteria. Preliminary studies have shown that some people at risk for ARDS have elevated ISGs in their neutrophils and that ISGs are associated with an impaired neutrophil response and increased severity of ARDS. This study will evaluate the association between viral-related neutrophil ISG response and the severity of ARDS.

Participants will include people on mechanical ventilation who are enrolled in either the ARDSNet 06 or 07 studies. For this study, participants will undergo blood collection within 48 hours of beginning the main ARDSNet study. There will be no study visits specifically for this study. Study researchers will analyze participants' blood samples and ARDSNet study data to gather information on mortality, the number of ventilator-free days, markers of severity of organ dysfunction and inflammation, and neutrophil response.

ELIGIBILITY:
Inclusion Criteria:

* All patients that are eligible for ARDSNet Study 06 (Prospective, Randomized, Multi-center Trial of Aerosolized Albuterol Versus Placebo in Patients with Acute Lung Injury [ALI] or Acute Respiratory Distress Syndrome [ARDS]) and ARDSNet Study 07 (Prospective, Randomized, Multi-center Trial of Initial Trophic Enteral Feeding Followed by Advancement to Full-Calorie Enteral Feeding vs. Early Advancement to Full-Calorie Enteral Feeding in Patients with Acute Lung Injury [ALI] or Acute Respiratory Distress Syndrome [ARDS] and Prospective, Randomized, Blinded, Placebo-controlled, Multi-center Trial of Omega-3 Fatty Acid, Gamma-Linolenic Acid, and Anti-Oxidant Supplementation in the Management of Acute Lung Injury [ALI] or Acute Respiratory Distress Syndrome [ARDS]) will be eligible for co-enrollment in this study
* Experiences acute onset of each of the following criteria within a 24-hour time period:

  1. Partial pressure of oxygen in arterial blood/fraction of inspired oxygen (PaO2/FiO2) less than or equal to 300; if altitude is greater than 1000 meters, then PaO2/FiO2 must be less than or equal to 300 x (barometric pressure [PB]/760)
  2. Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph. The infiltrates may be patchy, diffuse, homogeneous, or asymmetric.
  3. Requires positive pressure ventilation via endotracheal tube
  4. No clinical evidence of left-sided cardiac failure to account for bilateral pulmonary infiltrates

The 48-hour enrollment time window begins when the first three criteria are met. If a patient meets the first three inclusion criteria but has a pulmonary arterial wedge pressure (PAOP) greater than 18 mm Hg, then the first four criteria must persist for more than 12 hours after the PAOP has declined to less than or equal to 18 mm Hg, and still be within the 48-hour enrollment window.

Exclusion Criteria:

* More than 48 hours since all inclusion criteria were met
* Neuromuscular disease that impairs the ability to ventilate without assistance, such as cervical spinal cord injury at level C5 or higher, spinal cord injury, amyotrophic lateral sclerosis, Guillain-Barré syndrome, or myasthenia gravis
* Pregnant or breastfeeding
* Severe chronic respiratory disease, including chronic hypercapnia (arterial carbon dioxide pressure [PaCO2] greater than 45 mm Hg), chronic hypoxemia (PaO2 less than 55 mm Hg or FiO2 = 0.21), hospitalization within the 6 months prior to study entry for respiratory failure (PaCO2 greater than 50 mm Hg and/or PaO2 less than 55 mm Hg on 0.21 FiO2), secondary polycythemia, severe pulmonary hypertension (mean pulmonary arterial pressure [PAP] greater than 40 mm Hg), or ventilator dependency
* Burns over more than 40% of the total body surface area
* Cancer or other irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%
* Allogeneic bone marrow transplant within the 5 years prior to study entry
* Patient, surrogate, or physician is not committed to full support (exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)
* Severe chronic liver disease (i.e., Child-Pugh score between 11 and 15)
* Diffuse alveolar hemorrhage from vasculitis
* Morbid obesity (weighs greater than 1 kg/cm)
* Unwilling or unable to follow the ARDS network 6 mL/kg predicted body weight (PBW) ventilation protocol
* Not expected to survive 24 hours from the time of study entry
* No intent to obtain central venous access for monitoring intravascular pressures
* Medically unable to receive aerosolized albuterol
* Daily use (prior to study hospitalization) of inhaled beta agonist, corticosteroid, or oral leukotriene modifier
* Primary physician is unwilling to discontinue inpatient beta agonist use
* Acute heart attack or acute coronary syndrome within the 30 days prior to study entry
* Severe congestive heart failure
* Participation in other experimental medication trial in the 30 days prior to study entry with the exception of the ARDSNet pharmaconutrient nutrition trial (OMEGA)
* Heart rate greater than 85% of maximal predicted heart rate (MHR85) as calculated by MHR85 = 85% x (220-age)
* Receiving high frequency ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with Acute Lung Injury [ALI] or Acute Respiratory Distress Syndrome [ARDS] admitted to Intensive Care Units that are ARDSNet sites in Colorado.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2007-08; Primary Completion 2011-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure of subject mortality. | baseline to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A. Nick, MD, Principal Investigator — National Jewish Health
Locations (1):
- University of Colorado Health Sciences Center, Aurora, Colorado, United States

REFERENCES:
- [Background] Nick JA, Caceres SM, Kret JE, Poch KR, Strand M, Faino AV, Nichols DP, Saavedra MT, Taylor-Cousar JL, Geraci MW, Burnham EL, Fessler MB, Suratt BT, Abraham E, Moss M, Malcolm KC. Extremes of Interferon-Stimulated Gene Expression Associate with Worse Outcomes in the Acute Respiratory Distress Syndrome. PLoS One. 2016 Sep 8;11(9):e0162490. doi: 10.1371/journal.pone.0162490. eCollection 2016. PMID 27606687
- [Result] Malcolm KC, Kret JE, Young RL, Poch KR, Caceres SM, Douglas IS, Coldren CD, Burnham EL, Moss M, Nick JA. Bacteria-specific neutrophil dysfunction associated with interferon-stimulated gene expression in the acute respiratory distress syndrome. PLoS One. 2011;6(7):e21958. doi: 10.1371/journal.pone.0021958. Epub 2011 Jul 6. PMID 21755013